CLINICAL TRIAL: NCT00137787
Title: Randomized Controlled Trial Comparing Ciprofloxacin With Cefepime in Febrile Neutropenic Patients With Hematologic Diseases
Brief Title: Comparing Ciprofloxacin (CPFX) With Cefepime (CFPM) in Febrile Neutropenic Patients With Hematologic Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center for Supporting Hematology-Oncology Trials (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-SHOT 0402
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Febrile Neutropenia
Keywords: febrile neutropenia; hematologic disease
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Diseases | interventions — Ciprofloxacin; Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ciprofloxacin
- 2 (Active Comparator)
  Interventions: Drug: cefepime

INTERVENTIONS:
Drug: ciprofloxacin
  Arms: 1
Drug: cefepime
  Arms: 2

SUMMARY:
The aim of this study is to investigate whether intravenous ciprofloxacin is as effective as cefepime for the initial treatment of febrile neutropenia developed in patients with hematologic diseases.

DETAILED DESCRIPTION:
Infectious complications during neutropenic periods are major causes of morbidity and mortality especially for patients with hematological diseases, and prompt initiation of antibiotic therapy is warranted for those who develop febrile neutropenia. As for initial therapeutic agents, beta-lactam antibiotics, i.e., third- or fourth-generation cephalosporins and carbapenems have been used frequently because of their strong and broad-spectrum of action. However, under these conditions, development of resistance mediated by a beta-lactamase is concerned, and there is a need for alternative non-beta-lactam antibiotics for this indication. Ciprofloxacin is a potent agent covering against wide range of strains including Pseudomonas aeruginosa, and expected as a potential candidate. We have therefore planned a prospective randomized controlled trial designed to compare intravenous ciprofloxacin with cefepime for febrile neutropenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic disease
* Ages between 15 and 79 years
* Axillary temperature of 38.0 C or greater on one occasion or of 37.5 to 37.9 C lasting for more than 1 hour
* Absolute neutrophil count of less than 500/microL
* T-Bil level less than 2.0 times the upper limit of normal
* Cre level less than 1.5 times the upper limit of normal
* Written informed consent

Exclusion Criteria:

* Past history of allergic reaction to the study drug
* Positive for HIV antibody
* Pregnant or lactating women
* Family history of auditory disturbance
* Having received systemic antibacterial therapy within 14 days
* Receiving systemic antifungal or antiviral therapy except fluconazole or acyclovir for cases undergoing transplantation
* No recovery of neutrophil count of 1,000/microL or higher from the previous febrile episode
* On treatment with ketoprofen
* On treatment with sodium valproate
* Septic shock

Ages: 15 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | At 7 days after initiating therapy

SECONDARY OUTCOMES:
Treatment efficacy | At 21 days
Toxicity | During the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiko Atsuta, MD, Study Director — Nagoya University
Locations (1):
- Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- [Result] Yasuda T, Suzuki R, Ishikawa Y, Terakura S, Inamoto Y, Yanada M, Nagai H, Ozawa Y, Ozeki K, Atsuta Y, Emi N, Naoe T. Randomized controlled trial comparing ciprofloxacin and cefepime in febrile neutropenic patients with hematological malignancies. Int J Infect Dis. 2013 Jun;17(6):e385-90. doi: 10.1016/j.ijid.2012.12.005. Epub 2013 Jan 11. PMID 23317527